CLINICAL TRIAL: NCT04986865
Title: A First-in-Human Phase I Trial of ATG-101 in Patients With Metastatic/Advanced Solid Tumors and Mature B-cell Non-Hodgkin Lymphomas
Brief Title: A Study ATG-101 in Patients With Metastatic/Advanced Solid Tumors and Mature B-cell Non-Hodgkin Lymphomas
Acronym: PROBE
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: It is due to the recent changes in the competitor landscape and strategic consideration
Sponsor: Antengene Biologics Limited (Industry)
Responsible Party: Sponsor
Organization: Antengene Corporation (Industry)
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ATG-101-001
Record Dates: First submitted 2021-07-19; First posted 2021-08-03 (Actual); Last update posted 2025-06-09 (Actual); Status verified 2025-05

CONDITIONS: Advanced Solid Tumor; Metastatic Solid Tumor; Mature B-cell Non-Hodgkin Lymphoma
Keywords: Solid tumor, lymphoma, bispecific, antibody
MeSH Terms: conditions — Neoplasm Metastasis; Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Single experimental arm for ATG-101 (Experimental): Subjects with advanced or metastatic solid tumors and mature B-NHLs will be enrolled.
  Interventions: Drug: ATG-101

INTERVENTIONS:
Drug: ATG-101 — ATG-101 will be administered intravenously once every 21 days. During the Escalation Phase, the dose levels will be determined by the starting dose and the escalation steps taken in the trial. The Dose Expansion Phase will begin at the defined MTD, RP2D, or biologically optimal dose.

SUMMARY:
This is a First-in-Human Phase I trial of ATG-101 in Patients with Metastatic/Advanced Solid Tumors and Mature B-cell Non-Hodgkin Lymphomas.

DETAILED DESCRIPTION:
This is a First-in-Human Phase I trial of ATG-101 in Patients with Metastatic/Advanced Solid Tumors and Mature B-cell Non-Hodgkin Lymphomas. Dose Escalation Phase: Approximately 40-50 subjects with a maximum number of 62; Dose Expansion Phase: Estimated 100-400 subjects depending on the number of cohorts to be expanded.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated, written informed consent prior to any study-specific procedures, sampling, and analyses.
2. Aged at least 18 years as of the date of consent.
3. Histological or cytological confirmation of a solid tumor, and has progressed despite standard therapy, or is intolerant to standard therapy, or has a tumor for which no standard therapy exists or for which standard therapy is not considered adequate. Estimated life expectancy of a minimum of 12 weeks.
4. Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1.
5. Female and male subjects should be using adequate contraceptive measures as requested.

Exclusion Criteria:

1. Subjects with CNS tumors or known CNS metastases will be excluded.
2. Prior ATG-101 administration or a 4-1BB agonist.
3. Prior anti-tumor systemic therapy within 21 days(a period of 5 'half- lives') of the first dose of study treatment.
4. Radiotherapy with a wide field of radiation within 28 days.
5. With the exception of alopecia, any unresolved toxicities from prior therapy greater than Grade 1 (CTCAE v5.0) at the time of ICF signature.
6. Active infection, including hepatitis B and/or hepatitis C.
7. Have uncontrolled intercurrent illness, including but not limited to:
8. Inadequate bone marrow reserve or organ function.
9. History of hypersensitivity or history of allergic reactions attributed to drugs with a similar chemical or biologic structure or class to ATG-101.
10. Prior organ allograft transplantations.
11. Pregnant or nursing females.
12. Have a history of another primary malignancy within 3 years prior to starting study treatment. Exceptions are as follows: the disease under study; adequately treated basal or squamous cell carcinoma of the skin; cancer of the cervix in situ, etc.
13. In the opinion of the investigator, subject's complications or other conditions may affect protocol compliance or may be unsuitable for participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2021-12-15 (Actual); Primary Completion 2025-01-31 (Actual); Study Completion 2025-01-31 (Actual)

PRIMARY OUTCOMES:
AEs | One year after last patient first dose
  To evaluate the safety of ATG-101. It is the responsibility of the investigator to record and document all AEs (occurring from the first dose of study treatment on C1D1) throughout the study. Clinically significant symptoms and signs related to disease progression will be reported as AEs and meet one or more of the following criteria:
  1. With clinical symptoms.
  2. Leading to the change of study treatment (eg, dose adjustment, dose interruption, or study drug withdraw).
  3. Leading to the change of concomitant treatment (eg, adding, interrupting, or terminating concomitant medications, therapies, or treatments, or any other changes).
SAEs | One year after last patient first dose
  To evaluate the safety of ATG-101. It is the responsibility of the investigator to record and document all SAEs (occurring from the signing of the informed consent form) throughout the study. A SAE is any untoward medical occurrence that occurs at any dose (including SAEs occurred after the ICF is signed and prior to dosing):
  1. Results in death.
  2. Is life-threatening (immediate risk of death).
  3. Requires inpatient hospitalization or prolongation of existing hospitalization.
  4. Results in persistent or significant disability/incapacity.
  5. Is a congenital anomaly/birth defect. These should also usually be considered serious. Examples of such events are intensive treatment in an emergency room or at home for allergic bronchospasm, blood dyscrasias or convulsive that do not result in hospitalization; or development of drug dependency or drug abuse.
DLT (for Dose Escalation Phase only) | One year after last patient first dose
  The DLTs will be evaluated during Cycle 1 of treatment. Toxicity will be graded according to the National Cancer Institute-Common Terminology Criteria for Adverse Events. The DLTs for this study may include the following: Cytokine release syndrome, Hematologic toxicity, Non-hematologic toxicity.

SECONDARY OUTCOMES:
ORR | One year after last patient first dose
  To evaluate preliminary anti tumor activity of ATG-101
DOR | One year after last patient first dose
  To evaluate preliminary anti tumor activity of ATG-101
DCR | One year after last patient first dose
  To evaluate preliminary anti tumor activity of ATG-101
PFS | One year after last patient first dose
  To evaluate preliminary anti tumor activity of ATG-101
OS | One year after last patient first dose
  To evaluate preliminary anti tumor activity of ATG-101
The incidence of ADA and NAb | One year after last patient first dose
  To evaluate the immunogenicity of ATG-101
Serum concentrations of ATG-101 and derived PK parameters (for Dose Escalation Phase only) | One year after last patient first dose
  To characterize the PK of ATG 101 (for Dose Escalation Phase only)

CONTACTS AND LOCATIONS:
Locations (8):
- United States (3):
  - University of California San Francisco, San Francisco, California
  - Washington University School of Medicine in St. Louis, St Louis, Missouri
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
- Australia (5):
  - Scientia Clinical Research Ltd, Randwick, New South Wales
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Peter MacCallum Cancer Centre (PMCC) - Victorian Comprehensive Cancer Centre Location (Peter MacCallum Cancer Centre - East Melbourne), East Melbourne, Victoria
  - Austin Health - Olivia Newton-John Cancer Centre, Heidelberg, Victoria
  - The Alfred Hospital, Melbourne, Victoria